CLINICAL TRIAL: NCT05216328
Title: OMAMA-study - Prevention of Opioid-induced Constipation in Patients With Advanced Cancer
Brief Title: Prevention of Opioid-induced Constipation in Patients With Advanced Cancer
Acronym: OMAMA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Leiden University Medical Center (Other); University Medical Center Groningen (Other); Radboud University Medical Center (Other); Erasmus Medical Center (Other); Spaarne Gasthuis (Other); Rijnstate Hospital (Other); Jeroen Bosch Ziekenhuis (Other); Flevoziekenhuis (Other); Martini Hospital Groningen (Other); Haaglanden Medical Centre (Other); UMC Utrecht (Other); Groene Hart Ziekenhuis (Other); Bernhoven Hospital (Other); Isala (Other); Antoni van Leeuwenhoekziekenhuis (AVL) Amsterdam (Unknown)
Responsible Party: Principal Investigator, Lia van Zuylen, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08440012010002
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Constipation, Opioid-Induced
Keywords: Cancer; Palliative care; Cancer pain; Opioid-Induced Constipation; macrogol/electrolytes; magnesium hydroxide
MeSH Terms: conditions — Opioid-Induced Constipation; Neoplasms; Cancer Pain | interventions — Dosage Forms; Polyethylene Glycols; Electrolytes; Magnesium Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Macrogol/electrolytes (Active Comparator): Macrogol/electrolytes is started at a dose of 1 sachet once a day orally, based on the current guideline 'Diagnosis and treatment of pain in patients with cancer' (www.pallialine.nl). The dose of macrogol/electrolytes may be increased to 2 sachets a day during the study period.
  The effect of laxatives will be judged after 14 days.
  Interventions: Drug: Macrogol Only Product in Oral Dose Form
- Magnesium hydroxide (Active Comparator): Magnesium hydroxide is started at a dose of 724 mg three times a day orally, based on the current guideline 'Diagnosis and treatment of pain in patients with cancer' (www.pallialine.nl). The dose of magnesium hydroxide may be increased to 1448 mg three times a day during the study period. The effect of laxatives will be judged after 14 days.
  Interventions: Drug: Magnesium hydroxide 724mg

INTERVENTIONS:
Drug: Macrogol Only Product in Oral Dose Form — Information already included in arm/group description.
  Other Names: Macrogol/electrolytes
  Arms: Macrogol/electrolytes
Drug: Magnesium hydroxide 724mg — Information already included in arm/group description.
  Other Names: Magnesiumoxide
  Arms: Magnesium hydroxide

SUMMARY:
More than 70% of patients with cancer in the palliative phase have pain that often requires treatment with opioids (morphine-like agents). Constipation occurs in 59% of patients treated with opioids. Opioid-induced constipation (OIC) has consequences that range from daily discomfort with social insecurity and disability to intestinal obstruction. It leads to limitations in self-management, a reduced quality of life and a risk of the need for more care. In the guideline "Diagnosis and treatment of pain in patients with cancer" it is recommended to start preventively with an osmotic laxative such as macrogol/electrolytes or magnesium hydroxide when starting opioids. Macrogol/electrolytes has been proven to be effective for OIC, but is sometimes perceived by patients as unpleasant due to its taste. Magnesium hydroxide, which is less commonly prescribed for OIC, has a neutral taste. Although it is mentioned in the guideline, it is not studied for the treatment of OIC and also not officially registered for this. To support the advice of the guideline and to prove that a choice is possible, it is important to investigate whether there are differences in effectiveness and/or side effects between macrogol/electrolytes and magnesium hydroxide in the prevention of OIC.

The aim of this study is to compare macrogol/electrolytes with magnesium hydroxide in the prevention of opioid-induced constipation in patients with cancer in the palliative (incurable) phase, who start opioids because of pain. The choice of laxative is determined by drawing lots (randomisation). After two weeks, its effect will be assessed and will be presented as the percentage of patients who have not developed constipation after starting opioids. If the laxative, as assigned by lot, is described as satisfactory by the patient, the patient can continue with the drug that the patient used, after the study through regular prescription.

The investigators will ask the patients in the study about their satisfaction with the laxative used, any side effects and the degree of pain. Furthermore, the appeal to care for possible constipation will be examined. Because the best attainable quality of life in the palliative phase is the objective of all care, the investigators will also measure this perceived quality with a questionnaire in this study. The results of this study will lead to the best achievable prevention of opioid constipation in patients with cancer in the palliative phase.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Patients with metastatic cancer (≥18 years);
* Starting with slow release or transdermal opioids for pain;
* Able to complete a Dutch questionnaire. Previous treatment with opioids is allowed, if discontinued more than 4 weeks ago.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients with contra-indications for laxatives
* Use of laxatives during the last four weeks
* Severely impaired renal function (serum creatinine >180 umol/l)
* Estimated life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with a score of <30 of the Bowel Function Index | On day 14
  A clinician-administered patient-reported questionnaire to assess clinically significant constipation, validated in patients receiving opioids for chronic non-malignant pain and for malignant pain (Abramovitz 2013, Rentz 2009 and 2011). It consists of three questions, assessing ease of defecation, feeling of incomplete bowel evacuation and personal judgement of the patient regarding constipation, each during the last 7 days and each rated on a scale of 0 (best possible outcome) to 100 (worst possible outcome). A total score ≥30 (mean of the three separate scores) indicates clinically significant constipation. A change of the total score of >12 is regarded as clinically meaningful. It has been used in a large observational study in cancer patients receiving opioids (Davies 2021) and in randomised trials of opioid antagonists for OIC (Ahmedzai 2012, Dupoiron 2017, Leng 2020, Poelaert 2015). It has been recommended as the assessment tool of choice for OIC (Argoff 2015, Farmer 2019).

SECONDARY OUTCOMES:
The EQ5D | On day 0 and day 14
  A self-administered, generic assessment tool developed by the EuroQol Group, a network of international research teams, and consists of questions on five dimensions of health (i.e., mobility, self-care, pain/discomfort, usual activities, and anxiety/depression) (Pickard 2007). It has been used in cost-effectiveness studies on OIC (Dunlop 2012, Hjalte 2016, Lawson 2016).
Rome IV criteria for opioid-induced constipation | On day 0 and day 14
  Rome IV criteria for opioid-induced constipation as judged by professional care givers (Davies 2021, Drossman 2016), including:
  * straining during >25% of defecations
  * lumpy or hard stools in >25% of defecations
  * sensation of incomplete evacuation in >25% of defecations
  * sensation of anorectal obstruction/blockage in >25% of defecations
  * manual manoeuvres to facilitate >25% of defecations
  * <3 spontaneous defecations per week At least two of these criteria have to be fulfilled in order to diagnose constipation, to be judged by the treating physician or clinical nurse specialists/nurse practitioners
Cancer pain score | On day 0 and day 14
  Numeric Rating SDcale, ranging from 0 to 10
Patient satisfaction with laxative | On day 14
  A single four-item question, ranging from unsatisfied to very satisfied.
Side effects of laxatives | On day 14
  All side-effects are scored on a four-point Likert scale (not at all, a bit, rather, very much):
  * Bad taste
  * Problems with swallowing
  * Abdominal cramps
  * Nausea
  * Flatulence
  * Diarrhea
  * Other (to be specified by the patient)
Cost-effectiveness of macrogol/electrolytes compared to magnesium hydroxide | On day 14
  We aim to perform a comparative cost-effectiveness of the laxatives. This requires data collection on healthcare procedures and QOL in responders, non-responders and patients with side-effects of laxatives for the follow-up period of the study. These healthcare procedures will be extracted from hospital databases and healthcare use outside the hospital will be collected with the iMCQ at 4 weeks. All individual health care procedures will be linked to their unit costs. Reimbursement prices issued by the Dutch Healthcare Authority and national reference prices will be used for this assessment as outlined in current Dutch pharmaco-economic guidance. The cost-effectiveness analysis will be performed using a decision tree including different branches for initial therapy and responders and non-responders. The costs and QOL of the patients in the trial will be used as input for this decision tree. Total costs and effects will be calculated by summing the costs and effects of each branch.

CONTACTS AND LOCATIONS:
Overall Officials: Lia van Zuylen, Prof.dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (13):
- Netherlands (13):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - Radboud university Medical center Nijmegen, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Amsterdam UMC, location VUmc, Amsterdam, North Holland
  - Spaarne Gasthuis, Hoofddorp, North Holland
  - Groene Hart Hospital, Gouda, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haaglanden Medical Centre, The Hague, South Holland
  - University Medical Center Groningen, Groningen
  - Martini Hospital Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] Abramowitz L, Beziaud N, Causse C, Chuberre B, Allaert FA, Perrot S. Further validation of the psychometric properties of the Bowel Function Index for evaluating opioid-induced constipation (OIC). J Med Econ. 2013 Dec;16(12):1434-41. doi: 10.3111/13696998.2013.851083. Epub 2013 Oct 24. PMID 24102611
- [Background] Ahmedzai SH, Nauck F, Bar-Sela G, Bosse B, Leyendecker P, Hopp M. A randomized, double-blind, active-controlled, double-dummy, parallel-group study to determine the safety and efficacy of oxycodone/naloxone prolonged-release tablets in patients with moderate/severe, chronic cancer pain. Palliat Med. 2012 Jan;26(1):50-60. doi: 10.1177/0269216311418869. Epub 2011 Sep 21. PMID 21937568
- [Background] Argoff CE, Brennan MJ, Camilleri M, Davies A, Fudin J, Galluzzi KE, Gudin J, Lembo A, Stanos SP, Webster LR. Consensus Recommendations on Initiating Prescription Therapies for Opioid-Induced Constipation. Pain Med. 2015 Dec;16(12):2324-37. doi: 10.1111/pme.12937. Epub 2015 Nov 19. PMID 26582720
- [Background] Bell T, Annunziata K, Leslie JB. Opioid-induced constipation negatively impacts pain management, productivity, and health-related quality of life: findings from the National Health and Wellness Survey. J Opioid Manag. 2009 May-Jun;5(3):137-44. doi: 10.5055/jom.2009.0014. PMID 19662923
- [Background] Christensen HN, Olsson U, From J, Breivik H. Opioid-induced constipation, use of laxatives, and health-related quality of life. Scand J Pain. 2016 Apr;11:104-110. doi: 10.1016/j.sjpain.2015.12.007. Epub 2016 Jan 25. PMID 28850447
- [Background] Davies A, Leach C, Butler C, Gregory A, Henshaw S, Minton O, Shorthose K, Batsari KM. Opioid-induced constipation in patients with cancer: a "real-world," multicentre, observational study of diagnostic criteria and clinical features. Pain. 2021 Jan;162(1):309-318. doi: 10.1097/j.pain.0000000000002024. PMID 32701649
- [Background] Dhingra L, Shuk E, Grossman B, Strada A, Wald E, Portenoy A, Knotkova H, Portenoy R. A qualitative study to explore psychological distress and illness burden associated with opioid-induced constipation in cancer patients with advanced disease. Palliat Med. 2013 May;27(5):447-56. doi: 10.1177/0269216312450358. Epub 2012 Jun 15. PMID 22707180
- [Background] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Background] Dunlop W, Uhl R, Khan I, Taylor A, Barton G. Quality of life benefits and cost impact of prolonged release oxycodone/naloxone versus prolonged release oxycodone in patients with moderate-to-severe non-malignant pain and opioid-induced constipation: a UK cost-utility analysis. J Med Econ. 2012;15(3):564-75. doi: 10.3111/13696998.2012.665279. Epub 2012 Feb 23. PMID 22313329
- [Background] Dupoiron D, Stachowiak A, Loewenstein O, Ellery A, Kremers W, Bosse B, Hopp M. A phase III randomized controlled study on the efficacy and improved bowel function of prolonged-release (PR) oxycodone-naloxone (up to 160/80 mg daily) vs oxycodone PR. Eur J Pain. 2017 Oct;21(9):1528-1537. doi: 10.1002/ejp.1054. Epub 2017 Jun 22. PMID 28641363
- [Background] Farmer AD, Drewes AM, Chiarioni G, De Giorgio R, O'Brien T, Morlion B, Tack J. Pathophysiology and management of opioid-induced constipation: European expert consensus statement. United European Gastroenterol J. 2019 Feb;7(1):7-20. doi: 10.1177/2050640618818305. Epub 2018 Dec 14. PMID 30788113
- [Background] Freedman MD, Schwartz HJ, Roby R, Fleisher S. Tolerance and efficacy of polyethylene glycol 3350/electrolyte solution versus lactulose in relieving opiate induced constipation: a double-blinded placebo-controlled trial. J Clin Pharmacol. 1997 Oct;37(10):904-7. doi: 10.1002/j.1552-4604.1997.tb04264.x. PMID 9505981
- [Background] Ginex PK, Hanson BJ, LeFebvre KB, Lin Y, Moriarty KA, Maloney C, Vrabel M, Morgan RL. Management of Opioid-Induced and Non-Opioid-Related Constipation in Patients With Cancer: Systematic Review and Meta-Analysis. Oncol Nurs Forum. 2020 Nov 1;47(6):E211-E224. doi: 10.1188/20.ONF.E211-E224. PMID 33063777
- [Background] Hawley P, MacKenzie H, Gobbo M. PEG vs. sennosides for opioid-induced constipation in cancer care. Support Care Cancer. 2020 Apr;28(4):1775-1782. doi: 10.1007/s00520-019-04944-5. Epub 2019 Jul 18. PMID 31321524
- [Background] Head SJ, Kaul S, Bogers AJ, Kappetein AP. Non-inferiority study design: lessons to be learned from cardiovascular trials. Eur Heart J. 2012 Jun;33(11):1318-24. doi: 10.1093/eurheartj/ehs099. Epub 2012 May 7. PMID 22564354
- [Background] Hjalte F, Ragnarson Tennvall G, Welin KO, Westerling D. Treatment of Severe Pain and Opioid-induced Constipation: An Observational Study of Quality of Life, Resource Use, and Costs in Sweden. Pain Ther. 2016 Dec;5(2):227-236. doi: 10.1007/s40122-016-0059-9. Epub 2016 Nov 9. PMID 27830531
- [Background] Ishihara M, Ikesue H, Matsunaga H, Suemaru K, Kitaichi K, Suetsugu K, Oishi R, Sendo T, Araki H, Itoh Y; Japanese Study Group for the Relief of Opioid-induced Gastrointestinal Dysfunction. A multi-institutional study analyzing effect of prophylactic medication for prevention of opioid-induced gastrointestinal dysfunction. Clin J Pain. 2012 Jun;28(5):373-81. doi: 10.1097/AJP.0b013e318237d626. PMID 22156893
- [Background] Lyseng-Williamson KA. Correction to: Macrogol (polyethylene glycol) 4000 without electrolytes in the symptomatic treatment of chronic constipation: a profile of its use. Drugs Ther Perspect. 2019;35(1):49. doi: 10.1007/s40267-018-0588-x. Epub 2018 Nov 28. PMID 31186614
- [Background] Penning-van Beest FJ, van den Haak P, Klok RM, Prevoo YF, van der Peet DL, Herings RM. Quality of life in relation to constipation among opioid users. J Med Econ. 2010 Mar;13(1):129-35. doi: 10.3111/13696990903584436. PMID 20128662
- [Background] Pickard AS, Wilke CT, Lin HW, Lloyd A. Health utilities using the EQ-5D in studies of cancer. Pharmacoeconomics. 2007;25(5):365-84. doi: 10.2165/00019053-200725050-00002. PMID 17488136
- [Background] Poelaert J, Koopmans-Klein G, Dioh A, Louis F, Gorissen M, Loge D, Van Op den Bosch J, van Megen YJ. Treatment with prolonged-release oxycodone/naloxone improves pain relief and opioid-induced constipation compared with prolonged-release oxycodone in patients with chronic severe pain and laxative-refractory constipation. Clin Ther. 2015 Apr 1;37(4):784-92. doi: 10.1016/j.clinthera.2015.02.010. Epub 2015 Mar 7. PMID 25757607
- [Background] Rentz AM, Yu R, Muller-Lissner S, Leyendecker P. Validation of the Bowel Function Index to detect clinically meaningful changes in opioid-induced constipation. J Med Econ. 2009;12(4):371-83. doi: 10.3111/13696990903430481. PMID 19912069
- [Background] Rentz AM, van Hanswijck de Jonge P, Leyendecker P, Hopp M. Observational, nonintervention, multicenter study for validation of the Bowel Function Index for constipation in European countries. Curr Med Res Opin. 2011 Jan;27(1):35-44. doi: 10.1185/03007995.2010.535270. Epub 2010 Nov 18. PMID 21083515
- [Background] Taylor RR, Guest JF. The cost-effectiveness of macrogol 3350 compared to lactulose in the treatment of adults suffering from chronic constipation in the UK. Aliment Pharmacol Ther. 2010 Jan 15;31(2):302-12. doi: 10.1111/j.1365-2036.2009.04191.x. Epub 2009 Nov 3. PMID 19886948
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Tokoro A, Imai H, Fumita S, Harada T, Noriyuki T, Gamoh M, Akashi Y, Sato H, Kizawa Y. Incidence of opioid-induced constipation in Japanese patients with cancer pain: A prospective observational cohort study. Cancer Med. 2019 Aug;8(10):4883-4891. doi: 10.1002/cam4.2341. Epub 2019 Jun 24. PMID 31231974
- [Background] Wirz S, Klaschik E. Management of constipation in palliative care patients undergoing opioid therapy: is polyethylene glycol an option? Am J Hosp Palliat Care. 2005 Sep-Oct;22(5):375-81. doi: 10.1177/104990910502200511. PMID 16225360
- [Derived] Kistemaker KRJ, de Graeff A, Crul M, de Klerk G, van de Ven PM, van der Meulen MP, van Zuylen L, Steegers MAH. Magnesium hydroxide versus macrogol/electrolytes in the prevention of opioid-induced constipation in incurable cancer patients: study protocol for an open-label, randomized controlled trial (the OMAMA study). BMC Palliat Care. 2023 Mar 14;22(1):22. doi: 10.1186/s12904-023-01143-2. PMID 36915062
- See also: guidelines palliative care — http://www.pallialine.nl
- See also: The Dutch digital palliative care platform — http://www.palliaweb.nl